CLINICAL TRIAL: NCT00034164
Title: A Phase IIA Multicenter Evaluation of the Safety and Efficacy of Weekly Administration of S-8184 Paclitaxel Injectable Emulsion in Second Line Treatment of Patients With Relapsed Stage IIIB OR IV Non Small Cell Lung Cancer
Brief Title: Safety and Efficacy of S-8184 in Second Line Treatment of Relapsed Stage IIIB or IV Non Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Achieve Life Sciences (Industry)
Responsible Party: Monica Krieger, VP Regulatory Affairs, OncoGenex Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SON-8184-1063
Record Dates: First submitted 2002-04-23; First posted 2002-04-24 (Estimated); Last update posted 2009-06-04 (Estimated); Status verified 2009-06

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: S-8184 Paclitaxel Injectable Emulsion

SUMMARY:
Phase IIA, multicenter, dose escalation study evaluating the safety and efficacy of weekly S-8184 paclitaxel injectable emulsion in second line treatment of patients with relapsed stage IIIB or IV non small cell lung cancer.

DETAILED DESCRIPTION:
The goals of this study are to determine the objective response rate, to determine time to disease progression, duration of response, and survival, and to identify the maximum tolerated weekly dose and principal toxicities of S-8184 in this patient population.

ELIGIBILITY:
Inclusion Criteria:

Histologic diagnosis of non small cell lung cancer

Relapsed or unresectable stage IIIB or IV disease

One and only one prior cytotoxic chemotherapy regimen which must have included a platinum agent dosed at 60 mg/m2 or higher per cycle for cisplatin and AUC 6 per cycle for carboplatin

Documented response of at least stable disease while on first line therapy

Adult (18 years of age or older) patients

Adequate hematologic function (ANC greater than 1500 cells/mm3 and platelets greater than 100,000/mm3)

Serum creatinine less than 2.0 mg/dL

Total bilirubin less than 1.5 mg/dL; SGOT and SGPT less than 3 times the upper limit of institutional normal values

ECOG performance status of 0 - 2

Bidimensional measurable or clinically evaluable disease

Patients who have signed an IRB / Ethics Committee approved informed consent

Life expectancy at least 12 weeks

Patient has fully recovered from any previous surgery (at least 4 weeks since major surgery)

Patient has a negative pregnancy test prior to study entry if premenopausal. (Patients of child bearing potential must use a medically effective form of contraception during the treatment.)

Exclusion Criteria:

Patients who have received any taxane-containing preparation including Taxol (paclitaxel) or Taxotere (docetaxel)

Patients with intracranial metastases having neurologic function stabilized for less than 4 weeks prior to study entry

Females who are pregnant or lactating

Patients with peripheral neuropathy NCI-CTC grade 2 or greater

Patients who have received wide-field radiation, cytotoxic chemotherapy or hormonal therapy within 4 weeks of study entry; or mitomycin or nitrosoureas within 6 weeks of study entry

Patients who have had an investigational agent within 4 weeks of study entry

Patients receiving concurrent anticonvulsants known to induce P450 isoenzymes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2002-04; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
To determine the objective response rate | After all patients completed therapy

SECONDARY OUTCOMES:
To determine time to disease progression | After all patients completed therapy

CONTACTS AND LOCATIONS:
Locations (1):
- 3 Cities, Russia

REFERENCES:
- See also: sponsor's home page — http://www.sonuspharma.com